CLINICAL TRIAL: NCT04071327
Title: Pulmonary Hypertension Association Registry
Acronym: PHAR
Status: Recruiting | Type: Observational
Sponsor: Pulmonary Hypertension Association, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: PHAR
Record Dates: First submitted 2019-04-04; First posted 2019-08-28 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Arterial Hypertension; Chronic Thromboembolic Pulmonary Hypertension; Pulmonary Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pulmonary arterial hypertension (PAH): Patients with newly diagnosed or established PAH, within 6 months of first outpatient visit to a PH Care Center
- Chronic thromboembolic pulmonary hypertension (CTEPH): Patients with newly diagnosed or established CTEPH, within 6 months of first outpatient visit to a PH Care Center
- Group 3 PH due to Developmental Lung Disease: Pediatric patients with newly diagnosed or established Group 3 PH due to developmental lung disease, within 6 months of first outpatient visit to a PH Care Center.

SUMMARY:
The PHA Registry (PHAR) is a national study about people who have pulmonary arterial hypertension (PAH) and chronic thromboembolic pulmonary hypertension (CTEPH). PHAR collects information from people with PAH and CTEPH who are cared for in participating PHA-accredited Pulmonary Hypertension Care Centers throughout the U.S.

PHAR will determine how people with PAH and CTEPH are evaluated, tested, and treated, and will observe how well these participants do. The goal is to see if people with PH are treated according to recommended guidelines, and to see if there are certain factors that can lead to better or worse outcomes.

PHAR will include information about people with PAH and CTEPH in the U.S. who are seen at participating PHA-accredited PH Care Centers. PHAR contains data about patient care and outcomes. Specifically, data in the PHAR includes information on diagnosis; clinical status; socioeconomic status; diagnosis test results; body size; treatment information; interest in participating in clinical trials; family health and social history; and information about smoking, alcohol, or drug use. Participants are followed over time, and provide updates such as changes in therapy, how often participants need to go to the hospital, and survival. Such information may help healthcare providers provide better care.

ELIGIBILITY:
Inclusion Criteria:

* All age groups
* Written informed consent
* Pulmonary arterial hypertension (PAH), chronic thromboembolic pulmonary hypertension (CTEPH), or pediatric PH due to developmental lung disease
* Within 6 months of first outpatient visit at a PH Care Center

Exclusion Criteria:

* Diagnosis of WSPH Group 2 pulmonary hypertension
* Diagnosis of WSPH Group 3 pulmonary hypertension, except PH due to developmental lung disease
* Diagnosis of WSPH Group 5 pulmonary hypertension

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: New patients to a PHA-accredited PH Care Center (PHCC) with either newly diagnosed or established pulmonary arterial hypertension (PAH), chronic thromboembolic pulmonary hypertension (CTEPH), or pediatric PH due to developmental lung disease within 6 months of first outpatient visit at the PHCC.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2015-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of PAH and CTEPH patients completing all guideline-recommended diagnostics | 10 years
  PAH guideline-recommended diagnostics assessed include chest radiography, echocardiogram, ventilation-perfusion (V/Q) scan, pulmonary function tests, overnight oximetry, and right heart catheterization and identified as either "completed" or "not completed"
Impact of clinical predictors of disease worsening on patient outcomes | 10 years
  Prognostic importance of disease worsening predictors including changes in World Health Organization (WHO) / New York Heart Association (NYHA) functional class (I-IV), 6-minute walk distance in meters, and brain natriuretic peptide (BNP) in pg/mL on survival.
Survival | 10 years

CONTACTS AND LOCATIONS:
Locations (52):
- United States (52):
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - UC Davis Health, Sacramento, California
  - UCSF Medical Center, San Francisco, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Cottage Health System - Santa Barbara Pulmonary Associates, Santa Barbara, California
  - Stanford University, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - UC Health - Anschutz Medical Campus, Aurora, Colorado
  - University of Connecticut Health, Farmington, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - Northside Hospital, Atlanta, Georgia
  - Indiana University Health, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinic, Iowa City, Iowa
  - KU Medical Center, Kansas City, Kansas
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - Ochsner Medical Center, Jefferson, Louisiana
  - LSU Healthcare Network Clinic, New Orleans, Louisiana
  - University of MD Medical Group, PA, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota Health, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Weill Cornell Medical Center, New York, New York
  - Columbia University Medical Center/NewYork-Presbyterian Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - UNC Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - UC Health, Cincinnati, Ohio
  - The Oregon Clinic, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - Ft. Sanders Regional Medical Center, Knoxville, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Baylor Scott & White, Plano, Texas
  - University of Utah Health, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Heart Hospital, Norfolk, Virginia
  - VCU Medical Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hemnes AR, Beck GJ, Newman JH, Abidov A, Aldred MA, Barnard J, Berman Rosenzweig E, Borlaug BA, Chung WK, Comhair SAA, Erzurum SC, Frantz RP, Gray MP, Grunig G, Hassoun PM, Hill NS, Horn EM, Hu B, Lempel JK, Maron BA, Mathai SC, Olman MA, Rischard FP, Systrom DM, Tang WHW, Waxman AB, Xiao L, Yuan JX, Leopold JA; PVDOMICS Study Group. PVDOMICS: A Multi-Center Study to Improve Understanding of Pulmonary Vascular Disease Through Phenomics. Circ Res. 2017 Oct 27;121(10):1136-1139. doi: 10.1161/CIRCRESAHA.117.311737. PMID 29074534
- [Background] Tang WHW, Wilcox JD, Jacob MS, Rosenzweig EB, Borlaug BA, Frantz RP, Hassoun PM, Hemnes AR, Hill NS, Horn EM, Singh HS, Systrom DM, Tedford RJ, Vanderpool RR, Waxman AB, Xiao L, Leopold JA, Rischard FP. Comprehensive Diagnostic Evaluation of Cardiovascular Physiology in Patients With Pulmonary Vascular Disease: Insights From the PVDOMICS Program. Circ Heart Fail. 2020 Mar;13(3):e006363. doi: 10.1161/CIRCHEARTFAILURE.119.006363. Epub 2020 Feb 24. PMID 32088984
- [Background] Jellis CL, Park MM, Abidov A, Borlaug BA, Brittain EL, Frantz R, Hassoun PM, Horn EM, Jaber WA, Jiwon K, Karas MG, Kwon D, Leopold JA, Maron B, Mathai SC, Mehra R, Rischard F, Rosenzweig EB, Tang WHW, Vanderpool R, Thomas JD; PVDOMICS Study Group. Comprehensive echocardiographic evaluation of the right heart in patients with pulmonary vascular diseases: the PVDOMICS experience. Eur Heart J Cardiovasc Imaging. 2022 Jun 21;23(7):958-969. doi: 10.1093/ehjci/jeab065. PMID 34097027
- [Background] Hemnes AR, Leopold JA, Radeva MK, Beck GJ, Abidov A, Aldred MA, Barnard J, Rosenzweig EB, Borlaug BA, Chung WK, Comhair SAA, Desai AA, Dubrock HM, Erzurum SC, Finet JE, Frantz RP, Garcia JGN, Geraci MW, Gray MP, Grunig G, Hassoun PM, Highland KB, Hill NS, Hu B, Kwon DH, Jacob MS, Jellis CL, Larive AB, Lempel JK, Maron BA, Mathai SC, McCarthy K, Mehra R, Nawabit R, Newman JH, Olman MA, Park MM, Ramos JA, Renapurkar RD, Rischard FP, Sherer SG, Tang WHW, Thomas JD, Vanderpool RR, Waxman AB, Wilcox JD, Yuan JX, Horn EM; PVDOMICS Study Group. Clinical Characteristics and Transplant-Free Survival Across the Spectrum of Pulmonary Vascular Disease. J Am Coll Cardiol. 2022 Aug 16;80(7):697-718. doi: 10.1016/j.jacc.2022.05.038. PMID 35953136
- [Background] Frantz RP, Leopold JA, Hassoun PM, Hemnes AR, Horn EM, Mathai SC, Rischard FP, Larive AB, Tang WHW, Park MM, Hill NS, Rosenzweig EB. Acute vasoreactivity testing during right heart catheterization in chronic thromboembolic pulmonary hypertension: Results from the pulmonary vascular disease phenomics study. Pulm Circ. 2023 Jan 6;13(1):e12181. doi: 10.1002/pul2.12181. eCollection 2023 Jan. PMID 36618713
- [Background] Martens P, Yu S, Larive B, Borlaug BA, Erzurum SC, Farha S, Finet JE, Grunig G, Hemnes AR, Hill NS, Horn EM, Jacob M, Kwon DH, Park MM, Rischard FP, Rosenzweig EB, Wilcox JD, Tang WHW; PVDOMICS Study Group. Iron deficiency in pulmonary vascular disease: pathophysiological and clinical implications. Eur Heart J. 2023 Jun 9;44(22):1979-1991. doi: 10.1093/eurheartj/ehad149. PMID 36879444
- [Background] Simpson CE, Hemnes AR, Griffiths M, Grunig G, Tang WHW, Garcia JGN, Barnard J, Comhair SA, Damico RL, Mathai SC, Hassoun PM; PVDOMICS Study Group. Metabolomic Differences in Connective Tissue Disease-Associated Versus Idiopathic Pulmonary Arterial Hypertension in the PVDOMICS Cohort. Arthritis Rheumatol. 2023 Dec;75(12):2240-2251. doi: 10.1002/art.42632. Epub 2023 Oct 30. PMID 37335853
- [Background] Naranjo M, Rosenzweig EB, Hemnes AR, Jacob M, Desai A, Hill NS, Larive AB, Finet JE, Leopold J, Horn E, Frantz R, Rischard F, Erzurum S, Beck G, Mathai SC, Hassoun PM; PVDOMICS Study Group. Frequency of acute vasodilator response (AVR) in incident and prevalent patients with pulmonary arterial hypertension: Results from the pulmonary vascular disease phenomics study. Pulm Circ. 2023 Aug 21;13(3):e12281. doi: 10.1002/pul2.12281. eCollection 2023 Jul. PMID 37614830
- [Background] Simpson CE, Ambade AS, Harlan R, Roux A, Aja S, Graham D, Shah AA, Hummers LK, Hemnes AR, Leopold JA, Horn EM, Berman-Rosenzweig ES, Grunig G, Aldred MA, Barnard J, Comhair SAA, Tang WHW, Griffiths M, Rischard F, Frantz RP, Erzurum SC, Beck GJ, Hill NS, Mathai SC, Hassoun PM, Damico RL; the PVDOMICS Study Group. Kynurenine pathway metabolism evolves with development of preclinical and scleroderma-associated pulmonary arterial hypertension. Am J Physiol Lung Cell Mol Physiol. 2023 Nov 1;325(5):L617-L627. doi: 10.1152/ajplung.00177.2023. Epub 2023 Oct 3. PMID 37786941
- [Background] Lowery MM, Hill NS, Wang L, Rosenzweig EB, Bhat A, Erzurum S, Finet JE, Jellis CL, Kaur S, Kwon DH, Nawabit R, Radeva M, Beck GJ, Frantz RP, Hassoun PM, Hemnes AR, Horn EM, Leopold JA, Rischard FP, Mehra R; Pulmonary Vascular Disease Phenomics (PVDOMICS) Study Group. Sleep-Related Hypoxia, Right Ventricular Dysfunction, and Survival in Patients With Group 1 Pulmonary Arterial Hypertension. J Am Coll Cardiol. 2023 Nov 21;82(21):1989-2005. doi: 10.1016/j.jacc.2023.09.806. PMID 37968017
- [Background] Rischard FP, Bernardo RJ, Vanderpool RR, Kwon DH, Acharya T, Park MM, Katrynuik A, Insel M, Kubba S, Badagliacca R, Larive AB, Naeije R, Garcia JGN, Beck GJ, Erzurum SC, Frantz RP, Hassoun PM, Hemnes AR, Hill NS, Horn EM, Leopold JA, Rosenzweig EB, Tang WHW, Wilcox JD. Classification and Predictors of Right Ventricular Functional Recovery in Pulmonary Arterial Hypertension. Circ Heart Fail. 2023 Oct;16(10):e010555. doi: 10.1161/CIRCHEARTFAILURE.123.010555. Epub 2023 Sep 4. PMID 37664964
- [Derived] McCormick A, Krishnan A, Badesch D, Benza RL, Bull TM, De Marco T, Feldman J, Hemnes AR, Hirsch R, Horn E, Kennedy J, Mathai SC, McConnell W, Pugliese SC, Sager JS, Shlobin OA, Simon MA, Lammi MR. Pulmonary artery compliance in different forms of pulmonary hypertension. Heart. 2023 Jun 26;109(14):1098-1105. doi: 10.1136/heartjnl-2022-321760. PMID 36787969
- See also: Related Info — http://www.PHAssociation.org/PHAR